CLINICAL TRIAL: NCT05143879
Title: Long-term Effect of Combined Citrulline and Nitrate-rich Beetroot Extract Supplementation on Recovery Status in Trained Male Triathletes
Brief Title: Long-Term Effect of Combined Citrulline and Nitrate-Rich Beetroot Extract Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burgos Nutrition (Other)
Collaborators: Universidad de León (Other); University of the Basque Country (UPV/EHU) (Other); University of Valladolid (Other)
Responsible Party: Principal Investigator, Jose Burgos Balmaseda, Principal investigator, Burgos Nutrition
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ULE-020-2020
Record Dates: First submitted 2021-10-02; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Citrulline; Nitrate; Athletes
Keywords: triathlon; performance; ergogenic aids; muscle fatigue; recovery; hormones
MeSH Terms: interventions — Citrulline; Nitrates; Cellulose

STUDY DESIGN:
Intervention Model Description: The main purpose of this study was to determine the effect and degree of potentiation of the long-term (9 weeks) mixture of 3 g/day of CM plus 2.1 g/day of BEET (300 mg/day of NIT) supplementation on EIMD markers (urea, creatinine, AST, ALT, GGT, LDH and CK) and anabolic/catabolic hormone status (testosterone (T), cortisol (C), and T/C) in male trained triathletes.
Who Masked: Investigator
Masking Description: This study was a double-blind, placebo-controlled trial where participants (n = 32) were random-ized into 4 different groups: placebo group (PLG; n = 8), CIT group (CITG; 3 g/day of CIT; n = 8), BEET group (BEETG; 2.1 g/day of BEET (300 mg/day of NIT) ; n = 8) and CIT-NIT group (CIT-BEETG; 3 g/day of CIT plus 2.1 g/day of BEET (300 mg/day of NIT); n = 8)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): 8 subjects took 3 g/kg/day of placebo during 9 weeks
  Interventions: Dietary Supplement: Placebo
- Nitrate (Active Comparator): 8 subjects took 3 g/kg/day of nitrate during 9 weeks
  Interventions: Dietary Supplement: Nitrate
- Citrulline (Active Comparator): 8 subjects took 3 g/kg/day of citrulline during 9 weeks
  Interventions: Dietary Supplement: Citrulline
- Nitrate plus Citrulline (Active Comparator): 8 subjects took 3 g/kg/day of nitrate plus citrulline during 9 weeks
  Interventions: Dietary Supplement: Nitrate plus Citrulline

INTERVENTIONS:
Dietary Supplement: Citrulline — 3 g/day during 9 weeks
  Arms: Citrulline
Dietary Supplement: Nitrate — 300 mg/day during 9 weeks
  Arms: Nitrate
Dietary Supplement: Nitrate plus Citrulline — 3 g/day of citrulline and 300 mg/day of nitrate during 9 weeks
  Arms: Nitrate plus Citrulline
Dietary Supplement: Placebo — 3 g/day during 9 weeks
  Other Names: Cellulose
  Arms: Placebo

SUMMARY:
Citrulline (CIT) and nitrate-rich beetroot extract (BEET) are widely studied ergogenic aids. However, both supplements have been studied in sort-term and isolated. To the best of the authors' knowledge, the effects of combining both supplements on exercise-induced muscle damage (EIMD) and hormone status have not been investigated to date. Therefore, the main purpose of this study was to determine the effect and degree of potentiation of the long-term (9 weeks) mixture of 3 g/day of CIT plus 2.1 g/day of BEET (300 mg/day of NIT) supplementation on EIMD markers (urea, creatinine, AST, ALT, GGT, LDH and CK) and anabolic/catabolic hormone status (testosterone, cortisol and Testosterone cortisol ratio (T/C)) in male trained triathletes. This study was a double-blind, placebo-controlled trial where participants (n = 32) were randomized into 4 different groups: placebo group (PLG; n = 8), CIT group (CITG; 3 g/day of CIT; n = 8), BEET group (BEETG; 2.1 g/day of BEET (300 mg/day of NIT) ; n = 8) and CIT-NIT group (CIT-BEETG; 3 g/day of CIT plus 2.1 g/day of BEET (300 mg/day of NIT); n = 8). Blood samples were collected from all participants at baseline (T1) and after 9 weeks of supplementation (T2).

DETAILED DESCRIPTION:
Triathlon is an endurance sport in which athletes compete sequentially in swimming, cycling and running. Prolonged and strenuous training combined with insufficient recovery can produce muscular and metabolic stress, resulting in structural and functional damage to the musculoskeletal system leading to a fatigue status, which results in decreased athletic performance. As a consequence of this type of combined exercise, there are also alterations in biochemical markers of exercise-induced muscle damage (EIMD) as well as anabolic/catabolic hormones. Therefore, their analysis is useful in determining the balance between training loads and recovery. In this sense, it is essential to include different strategies to reduce or prevent EIMD, which delay or reduce muscle fatigue and improve sports performance. One of these strategies is the use of different ergogenic aids such as L-citrulline (CIT) and nitrates (NIT) which have been proposed as both substances produce an increase in nitric oxide (NO).

ELIGIBILITY:
Inclusion Criteria:

* Males between 25 and 35 years old
* Triathletes
* With at least 5 years of experience
* Without any disease
* Non smokers
* Non drinkers of alcohol
* Not to take any other medications or stimulant substances during the study
* 2 weeks without taking other nutritional supplements

Exclusion Criteria:

* Exclusion criteria:
* Men under 25 and over 35 years of age.
* Non triathletes
* Less than 5 years of experience
* With any disease
* Smokers
* Alcohol drinkers

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Cortisol | 9 weeks
  μg/dL
Testosterone | 9 weeks
  ng/mL
Testosterone to cortisol ratio | 9 weeks
  ng/mL
Urea | 9 weeks
  mg/dl
Creatinine | 9 weeks
  mg/dl
AST | 9 weeks
  U/L
ALT | 9 weeks
  U/L
GGT | 9 weeks
  U/L
LDH | 9 weeks
  U/L
CK | 9 weeks
  U/L

CONTACTS AND LOCATIONS:
Overall Officials: Jose Burgos Balmaseda, Graduate, Principal Investigator — University of Leon
Locations (1):
- University of Leon, León, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gonzalez AM, Trexler ET. Effects of Citrulline Supplementation on Exercise Performance in Humans: A Review of the Current Literature. J Strength Cond Res. 2020 May;34(5):1480-1495. doi: 10.1519/JSC.0000000000003426. PMID 31977835
- [Result] Gilligan DM, Panza JA, Kilcoyne CM, Waclawiw MA, Casino PR, Quyyumi AA. Contribution of endothelium-derived nitric oxide to exercise-induced vasodilation. Circulation. 1994 Dec;90(6):2853-8. doi: 10.1161/01.cir.90.6.2853. PMID 7994830
- [Result] Anderson JE. A role for nitric oxide in muscle repair: nitric oxide-mediated activation of muscle satellite cells. Mol Biol Cell. 2000 May;11(5):1859-74. doi: 10.1091/mbc.11.5.1859. PMID 10793157
- [Result] Bailey SJ, Blackwell JR, Lord T, Vanhatalo A, Winyard PG, Jones AM. l-Citrulline supplementation improves O2 uptake kinetics and high-intensity exercise performance in humans. J Appl Physiol (1985). 2015 Aug 15;119(4):385-95. doi: 10.1152/japplphysiol.00192.2014. Epub 2015 May 28. PMID 26023227
- [Result] Viribay A, Arribalzaga S, Mielgo-Ayuso J, Castaneda-Babarro A, Seco-Calvo J, Urdampilleta A. Effects of 120 g/h of Carbohydrates Intake during a Mountain Marathon on Exercise-Induced Muscle Damage in Elite Runners. Nutrients. 2020 May 11;12(5):1367. doi: 10.3390/nu12051367. PMID 32403259
- [Result] Wang JM, Gu CH, Tao L, Wu XL. Effect of surgery and efferent duct ligation on testicular blood flow and testicular steroidogenesis in the rat. J Reprod Fertil. 1985 Jan;73(1):191-6. doi: 10.1530/jrf.0.0730191. PMID 3968652
- [Result] Monau TR, Vargas VE, Zhang L, Myers DA, Ducsay CA. Nitric oxide inhibits ACTH-induced cortisol production in near-term, long-term hypoxic ovine fetal adrenocortical cells. Reprod Sci. 2010 Oct;17(10):955-62. doi: 10.1177/1933719110376092. Epub 2010 Aug 16. PMID 20713972
- [Result] Milton-Laskibar I, Martinez JA, Portillo MP. Current Knowledge on Beetroot Bioactive Compounds: Role of Nitrate and Betalains in Health and Disease. Foods. 2021 Jun 7;10(6):1314. doi: 10.3390/foods10061314. PMID 34200431
- [Result] Clifford T, Bell O, West DJ, Howatson G, Stevenson EJ. The effects of beetroot juice supplementation on indices of muscle damage following eccentric exercise. Eur J Appl Physiol. 2016 Feb;116(2):353-62. doi: 10.1007/s00421-015-3290-x. Epub 2015 Nov 4. PMID 26537365
- [Result] Garnacho-Castano MV, Palau-Salva G, Serra-Paya N, Ruiz-Hermosel M, Berbell M, Vinals X, Bataller MG, Carbonell T, Vilches-Saez S, Cobo EP, Molina-Raya L. Understanding the effects of beetroot juice intake on CrossFit performance by assessing hormonal, metabolic and mechanical response: a randomized, double-blind, crossover design. J Int Soc Sports Nutr. 2020 Nov 13;17(1):56. doi: 10.1186/s12970-020-00388-z. PMID 33187518
- [Result] da Silva DK, Jacinto JL, de Andrade WB, Roveratti MC, Estoche JM, Balvedi MCW, de Oliveira DB, da Silva RA, Aguiar AF. Citrulline Malate Does Not Improve Muscle Recovery after Resistance Exercise in Untrained Young Adult Men. Nutrients. 2017 Oct 18;9(10):1132. doi: 10.3390/nu9101132. PMID 29057836
- [Result] Wax B, Kavazis AN, Luckett W. Effects of Supplemental Citrulline-Malate Ingestion on Blood Lactate, Cardiovascular Dynamics, and Resistance Exercise Performance in Trained Males. J Diet Suppl. 2016;13(3):269-82. doi: 10.3109/19390211.2015.1008615. Epub 2015 Feb 12. PMID 25674699
- [Result] Perez-Guisado J, Jakeman PM. Citrulline malate enhances athletic anaerobic performance and relieves muscle soreness. J Strength Cond Res. 2010 May;24(5):1215-22. doi: 10.1519/JSC.0b013e3181cb28e0. PMID 20386132
- [Result] McMahon NF, Leveritt MD, Pavey TG. The Effect of Dietary Nitrate Supplementation on Endurance Exercise Performance in Healthy Adults: A Systematic Review and Meta-Analysis. Sports Med. 2017 Apr;47(4):735-756. doi: 10.1007/s40279-016-0617-7. PMID 27600147
- [Result] Jones AM, Thompson C, Wylie LJ, Vanhatalo A. Dietary Nitrate and Physical Performance. Annu Rev Nutr. 2018 Aug 21;38:303-328. doi: 10.1146/annurev-nutr-082117-051622. PMID 30130468
- [Result] Richards JC, Racine ML, Hearon CM Jr, Kunkel M, Luckasen GJ, Larson DG, Allen JD, Dinenno FA. Acute ingestion of dietary nitrate increases muscle blood flow via local vasodilation during handgrip exercise in young adults. Physiol Rep. 2018 Jan;6(2):e13572. doi: 10.14814/phy2.13572. PMID 29380952
- [Result] Curis E, Nicolis I, Moinard C, Osowska S, Zerrouk N, Benazeth S, Cynober L. Almost all about citrulline in mammals. Amino Acids. 2005 Nov;29(3):177-205. doi: 10.1007/s00726-005-0235-4. Epub 2005 Aug 8. PMID 16082501
- [Result] Rammos C, Luedike P, Hendgen-Cotta U, Rassaf T. Potential of dietary nitrate in angiogenesis. World J Cardiol. 2015 Oct 26;7(10):652-7. doi: 10.4330/wjc.v7.i10.652. PMID 26516419
- [Result] Wylie LJ, Park JW, Vanhatalo A, Kadach S, Black MI, Stoyanov Z, Schechter AN, Jones AM, Piknova B. Human skeletal muscle nitrate store: influence of dietary nitrate supplementation and exercise. J Physiol. 2019 Dec;597(23):5565-5576. doi: 10.1113/JP278076. Epub 2019 Jul 27. PMID 31350908
- [Result] Daab W, Bouzid MA, Lajri M, Bouchiba M, Saafi MA, Rebai H. Chronic Beetroot Juice Supplementation Accelerates Recovery Kinetics following Simulated Match Play in Soccer Players. J Am Coll Nutr. 2021 Jan;40(1):61-69. doi: 10.1080/07315724.2020.1735571. Epub 2020 Mar 3. PMID 32125249